CLINICAL TRIAL: NCT03246620
Title: Oro-dispersible Olanzapine (Wafer) Versus Conventional Oral Haloperidol or Diazepam Tablets for the Management of Acute Agitation in the Accident and Emergency Department - a Multicentre Randomised Clinical Trial
Brief Title: Oral Olanzapine Versus Haloperidol or Diazepam
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated prematurely due to difficulties in patient recruitment and associated potential for selection bias.
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Esther Wai Yin Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChanEW oral sedation RCT; 17111615 (Other Grant/Funding Number: Research Grant Council, Hong Kong)
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Acute Agitation; Behavioural Emergency
Keywords: emergency; emergency medicine; sedation; acute agitation
MeSH Terms: conditions — Emergencies | interventions — Olanzapine; Haloperidol; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Olanzapine (Experimental): oro-dispersible tablet (wafer)(Zyprexa), 5 mg, single dose
  Interventions: Drug: Olanzapine oro-dispersible 5Mg Tab
- Haloperidol (Active Comparator): Haloperidol encapsulated tablet, 2 mg tablet, single dose
  Interventions: Drug: Haloperidol 2Mg encapsulated Tab
- Diazepam (Active Comparator): Diazepam encapsulated tablet, 2mg tablet, single dose
  Interventions: Drug: Diazepam 2Mg encapsulated Tab

INTERVENTIONS:
Drug: Olanzapine oro-dispersible 5Mg Tab — Patient allocated to this arm will be given 5 mg olanzapine oro-dispersible tablet and an encapsulated placebo tablet
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Haloperidol 2Mg encapsulated Tab — Patient allocated to this arm will be given 2 mg encapsulated haloperidol tablet and an oro-dispersible placebo tablet
  Arms: Haloperidol
Drug: Diazepam 2Mg encapsulated Tab — Patient allocated to this arm will be given 2 mg encapsulated diazepam tablet and an oro-dispersible placebo tablet
  Arms: Diazepam

SUMMARY:
The purpose of this study is to determine whether oral olanzapine is safer (fewer adverse events) and more effective (shorter time to sedation) than conventional haloperidol or diazepam when used in the management of acute agitation in the emergency.

DETAILED DESCRIPTION:
1. Investigate oral use of sedating drugs within a predominantly Chinese population, to address this void in international literature impacting the management of acute agitation.
2. The multi-centre Randomised Clinical Trial will determine the safety and efficacy of oral olanzapine, in comparison with conventional medicines (haloperidol or diazepam) in a three-arm comparison for the sedation of acutely agitated patients in AEDs. Specifically, we aim to determine if administration of oral olanzapine (a)is more effective than sedation with oral haloperidol or oral diazepam alone; (b)is safer than sedation with comparison arms; (c)decreases the amount of subsequent redosing or alternative drugs required; (d)is more favourable than the haloperidol and diazepam arms with respect to safety, efficacy and adverse events.

Investigate potential variables leading to AED attendance and/or admission requiring oral sedation. These may include patient demographic and regular medications and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Accident & Emergency Department patients
* Requiring oral drug sedation (as determined by an emergency clinician) will be enrolled.

Exclusion Criteria:

* known hypersensitivity or contraindication to the study drugs
* reversible aetiology for agitation (e.g. hypotension, hypoxia, hypoglycaemia)
* known pregnancy
* acute alcohol withdrawal
* refusal to take oral medication
* patients from correctional facilities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Time to achieve adequate sedation | Within 60 minutes from drug administration
  Adequate sedation is determined by a 6-point validated scale

SECONDARY OUTCOMES:
Total study drug doses administered; alternative drugs and doses used | From Accident & Emergency Department(AED) admission to transfer or discharge from AED, an expected average of 1 hour
Corrected QT interval (QTc) | From Accident & Emergency Department(AED) admission to transfer or discharge from AED, an expected average of 1 hour
AED length of stay (LOS) | From Accident & Emergency Department(AED) admission to transfer or discharge from AED, an expected average of 1 hour
Adverse events | From Accident & Emergency Department(AED) admission to transfer or discharge from AED, an expected average of 1 hour
  including airway management (jaw thrust, oral, nasal airway), need for assisted ventilation (bag/mask, intubation), oxygen desaturation <90%, systolic BP<90 mmHg, dystonic reactions, seizures, vomiting or aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Knott JC, Bennett D, Rawet J, Taylor DM. Epidemiology of unarmed threats in the emergency department. Emerg Med Australas. 2005 Aug;17(4):351-8. doi: 10.1111/j.1742-6723.2005.00756.x. PMID 16091097
- [Background] Chan EW, Taylor DM, Knott JC, Phillips GA, Castle DJ, Kong DC. Intravenous droperidol or olanzapine as an adjunct to midazolam for the acutely agitated patient: a multicenter, randomized, double-blind, placebo-controlled clinical trial. Ann Emerg Med. 2013 Jan;61(1):72-81. doi: 10.1016/j.annemergmed.2012.07.118. Epub 2012 Sep 13. PMID 22981685
- [Background] Knott JC, Taylor DM, Castle DJ. Randomized clinical trial comparing intravenous midazolam and droperidol for sedation of the acutely agitated patient in the emergency department. Ann Emerg Med. 2006 Jan;47(1):61-7. doi: 10.1016/j.annemergmed.2005.07.003. Epub 2005 Aug 18. PMID 16387219
- [Background] Chan EW, Taylor DM, Knott JC, Kong DC. Variation in the management of hypothetical cases of acute agitation in Australasian emergency departments. Emerg Med Australas. 2011 Feb;23(1):23-32. doi: 10.1111/j.1742-6723.2010.01348.x. Epub 2010 Nov 22. PMID 21091874
- [Background] Chan EW, Knott JC, Taylor DM, Phillips GA, Kong DC. Intravenous olanzapine--another option for the acutely agitated patient? Emerg Med Australas. 2009 Jun;21(3):241-2. doi: 10.1111/j.1742-6723.2009.01190.x. No abstract available. PMID 19527287
- [Background] Chan EW, Taylor DM, Knott JC, Liew D, Kong DC. The pharmacoeconomics of managing acute agitation in the emergency department: what do we know and how do we approach it? Expert Rev Pharmacoecon Outcomes Res. 2012 Oct;12(5):589-95. doi: 10.1586/erp.12.53. PMID 23186399
- [Background] Chan EW, Tang C, Lao KS, Ling Pong L, Tsui MS, Ho HF, Wong GC, Kong DC, McD Taylor D, Knott JC, Wong IC. Management of acute agitation in Hong Kong and comparisons with Australasia. Emerg Med Australas. 2015 Dec;27(6):542-548. doi: 10.1111/1742-6723.12499. Epub 2015 Dec 3. PMID 26635127
- [Background] Yap CYL, Taylor DM, Knott JC, Taylor SE, Phillips GA, Karro J, Chan EW, Kong DCM, Castle DJ. Intravenous midazolam-droperidol combination, droperidol or olanzapine monotherapy for methamphetamine-related acute agitation: subgroup analysis of a randomized controlled trial. Addiction. 2017 Jul;112(7):1262-1269. doi: 10.1111/add.13780. Epub 2017 Feb 28. PMID 28160494